CLINICAL TRIAL: NCT00406614
Title: Health Literacy Intervention for Korean Americans With High Blood Pressure (HBP)
Brief Title: Health Literacy-Focused Program to Improve Blood Pressure Control in Korean Americans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Miyong Kim, Professor, Johns Hopkins University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 446; R01HL085567 (NIH)
Record Dates: First submitted 2006-11-30; First posted 2006-12-04 (Estimated); Last update posted 2017-03-08 (Actual); Status verified 2011-11

CONDITIONS: Hypertension
Keywords: High Blood Pressure
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Literacy-focused high blood pressure intervention. The intervention group will receive the health literacy -focused hypertension management intervention that will be delivered through 6 weeks of highly interactive group sessions in a classroom setting, followed by telephone counseling once a month for 12 months. Also, the intervention group will concurrently use home blood pressure monitoring with telephone transmission for 12 months.
  Interventions: Behavioral: Health Literacy-Focused High Blood Pressure Intervention
- 2 (Active Comparator): Wait-list control group will initially receive usual care from a regular medical provider. Participants in the control group will take part in the intervention once the study has been completed.
  Interventions: Behavioral: Health Literacy-Focused High Blood Pressure Intervention

INTERVENTIONS:
Behavioral: Health Literacy-Focused High Blood Pressure Intervention — Participants assigned to the intervention group will attend a weekly 2-hour educational session for 6 weeks that will cover topics such as learning medical terminology, understanding the content of prescription and appointment slips, and blood pressure (BP) management strategies. Upon completion of the educational sessions, participants will submit BP measurements via telephone monitoring system for 12 months and Community Health Worker (CHW) will conduct telephone counseling once every month during the same 12-month period for support and follow-up counseling. Participants will continue to monitor BP measurement by logging BP data on BP diary book for another 12 months. Control group participants will receive the same intervention education following the completion of the study.
  Other Names: SI - intervention receiving group

SUMMARY:
Many Korean Americans are at risk for developing high blood pressure. Low health literacy levels may play a role in this risk. The purpose of this study is to evaluate a literacy-focused program aimed at reducing blood pressure levels in older Korean Americans.

DETAILED DESCRIPTION:
In the last decade, significant progress has been made in improving the heart health of individuals in the United States. However, despite these advances, many racial and ethnic minority groups still have high rates of cardiovascular disease. Korean Americans, in particular, are more prone to developing high blood pressure than other Americans or individuals living in Korea. Possible reasons for this may include stress, diet, or lifestyle changes that occur as a result of immigration. Because many Korean Americans have low health literacy skills, it may be harder for them to understand medication dosing instructions, keep track of medical appointments, or comprehend written medical information. Korean Americans have traditionally been identified as a "hard to reach" group, and few programs have specifically targeted these individuals with regards to improving blood pressure control. The purpose of this study is to evaluate a health literacy-focused intervention that aims to improve blood pressure control among older Korean Americans. The results from this study may be helpful in developing future literacy-focused blood pressure programs targeted to minority groups in the United States.

In this study, participants will be randomly assigned to either a literacy-focused high blood pressure intervention or a wait-list control group, which will initially involve usual care from a regular medical provider. Participants in the intervention group will attend a weekly 2-hour educational session for 6 weeks. Bilingual research nurses and other professionals will facilitate these sessions, and each participant will receive a Korean language workbook with examples of medical terminology, prescription and appointment slips, and blood pressure management strategies. For 12 months, participants will self-monitor their blood pressure and record these measurements through a telephone management system. Community health workers will conduct telephone counseling on a monthly basis and those participants with uncontrolled blood pressure will receive more intensive support and follow-up counseling. Study visits will occur at Week 6 and Months 6, 12, 18, and 24, at which time blood pressure, height, and weight will be measured. In addition, participants will complete questionnaires that assess health literacy, high blood pressure knowledge, problem solving and communication skills, treatment adherence, health care utilization, and quality of life. Participants in the control group will take part in the intervention once the study has been completed.

ELIGIBILITY:
Inclusion Criteria:

* Self-identifies as a first-generation Korean American
* Systolic blood pressure greater than 140 mm Hg and/or diastolic blood pressure greater than 90 mm Hg OR currently on medication to treat high blood pressure
* Access to a telephone

Exclusion Criteria:

* Current participation in another clinical trial
* Acute and/or terminal medical condition that would make study participation difficult (e.g., terminal cancer, acute heart attack)
* Psychiatric diagnosis that would make study participation difficult (e.g., schizophrenia, cognitive impairment)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2007-09; Primary Completion 2009-08 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Health literacy levels | Measured at Week 6 and Months 6, 12, 18, and 24
Blood pressure control | Measured at Week 6 and Months 6, 12, 18, and 24
Reduction in blood pressure | Measured at Month 24

SECONDARY OUTCOMES:
High blood pressure knowledge | Measured at Week 6 and Months 6, 12, 18, and 24
Problem solving and communication skills | Measured at Week 6 and Months 6, 12, 18, and 24
Adherence to high blood pressure treatment recommendations | Measured at Week 6 and Months 6, 12, 18, and 24
Health care utilization | Measured at Week 6 and Months 6, 12, 18, and 24
High blood pressure-related quality of life | Measured at Month 24

CONTACTS AND LOCATIONS:
Overall Officials: Miyong T. Kim, PhD, Principal Investigator — The Johns Hopkins University School of Nursing
Locations (1):
- Korean Resource Center, Ellicott City, Maryland, United States

REFERENCES:
- [Derived] Kim MT, Kim KB, Han HR, Huh B, Nguyen T, Lee HB. Prevalence and Predictors of Depression in Korean American Elderly: Findings from the Memory and Aging Study of Koreans (MASK). Am J Geriatr Psychiatry. 2015 Jul;23(7):671-83. doi: 10.1016/j.jagp.2014.11.003. Epub 2014 Nov 25. PMID 25554484
- [Derived] Kim KB, Han HR, Huh B, Nguyen T, Lee H, Kim MT. The effect of a community-based self-help multimodal behavioral intervention in Korean American seniors with high blood pressure. Am J Hypertens. 2014 Sep;27(9):1199-208. doi: 10.1093/ajh/hpu041. Epub 2014 Mar 26. PMID 24671049
- [Derived] Lee JE, Kim MT, Han HR. Correlates of Health-Related Quality of Life Among Korean Immigrant Elders. J Appl Gerontol. 2015 Oct;34(7):844-57. doi: 10.1177/0733464813490247. Epub 2013 Jun 11. PMID 24652887
- [Derived] Han HR, Park SY, Song H, Kim M, Kim KB, Lee HB. Feasibility and validity of dementia assessment by trained community health workers based on Clinical Dementia Rating. J Am Geriatr Soc. 2013 Jul;61(7):1141-5. doi: 10.1111/jgs.12309. Epub 2013 Jun 3. PMID 23730928
- [Derived] Han HR, Song Y, Song HJ, Kim MT. Influence of living arrangements on the management and control of hypertension: a mixed-methods study of Korean American elderly. J Immigr Minor Health. 2013 Oct;15(5):944-52. doi: 10.1007/s10903-012-9679-2. PMID 22790881
- [Derived] Kim MT, Song HJ, Han HR, Song Y, Nam S, Nguyen TH, Lee HC, Kim KB. Development and validation of the high blood pressure-focused health literacy scale. Patient Educ Couns. 2012 May;87(2):165-70. doi: 10.1016/j.pec.2011.09.005. Epub 2011 Oct 24. PMID 22030252
- [Derived] Han HR, Chan K, Song H, Nguyen T, Lee JE, Kim MT. Development and evaluation of a hypertension knowledge test for Korean hypertensive patients. J Clin Hypertens (Greenwich). 2011 Oct;13(10):750-7. doi: 10.1111/j.1751-7176.2011.00497.x. Epub 2011 Jul 14. PMID 21974763
- See also: Click here for the Korean Resource Center web site — http://www.ikorean.org/